CLINICAL TRIAL: NCT07381504
Title: Acute Aerobic Exercise Intervention for Children With Autism Spectrum Disorder and Co-Occurring Sleep Disorder
Brief Title: Aerobic Exercise for Sleep in Children With ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202407160RINE
Record Dates: First submitted 2025-12-28; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Sleep Disorders; Acute Aerobic Exercise; Physical Fitness; Children
MeSH Terms: conditions — Autism Spectrum Disorder; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic-Cognitive Behavioral Integrated Intervention (ACBI) program (Experimental): The Aerobic-Cognitive Behavioral Integrated Intervention (ACBI) combines supervised moderate-to-vigorous aerobic exercise (twice weekly, 30 minutes per session for 2 weeks) with a parent-mediated cognitive behavioral component targeting sleep-related behaviors. Exercise intensity is monitored using heart rate-based criteria. Parents receive structured guidance and implement cognitive behavioral strategies daily at home throughout the intervention period.
  Interventions: Behavioral: Intervention 1: Acute Aerobic Exercise; Behavioral: Intervention 2: Parent-Mediated Cognitive Behavioral Training
- Control group (Active Comparator): Provision of written materials describing cognitive behavioral strategies for managing sleep-related behaviors in children with ASD. No structured training sessions or supervised implementation are provided.
  Interventions: Behavioral: Parent Self-Education Program

INTERVENTIONS:
Behavioral: Intervention 1: Acute Aerobic Exercise — Moderate-to-vigorous-intensity intermittent aerobic exercise conducted twice per week, 30 minutes per session, over a 2-week period. Exercise intensity is prescribed and monitored using heart rate-based criteria. All sessions are supervised by trained research staff.
  Arms: Aerobic-Cognitive Behavioral Integrated Intervention (ACBI) program
Behavioral: Intervention 2: Parent-Mediated Cognitive Behavioral Training — Structured parent training in cognitive behavioral strategies targeting sleep-related behaviors, including sleep routines, environmental modifications, and behavioral reinforcement techniques. Parents are instructed to implement strategies daily at home throughout the intervention period.
  Arms: Aerobic-Cognitive Behavioral Integrated Intervention (ACBI) program
Behavioral: Parent Self-Education Program — Children with ASD in the control group were provided with a Cognitive Behavioral Strategy Information, in which parents received written materials describing cognitive behavioral strategies relevant to supporting children's self-regulation and daily behaviors. Parents were encouraged to review the materials and apply the strategies at home as they deemed appropriate. No structured training sessions or supervised implementation were provided.
  Arms: Control group

SUMMARY:
Autism Spectrum Disorder (ASD) is a neurodevelopmental condition characterized by impairments in social interaction and communication. Children with ASD frequently experience co-occurring behavioral problems, among which sleep disturbances are highly prevalent, affecting approximately 40%-80% of children and adolescents with ASD. These sleep problems pose a substantial burden during childhood and adolescence.

This study employs a two-phase design to examine the effects of an acute aerobic exercise intervention combined with a parent-mediated cognitive behavioral program on sleep problems in children with autism spectrum disorder (ASD). Phase 1 consists of cross-sectional assessments comparing sleep efficiency, physical fitness, and attentional performance among children with ASD with and without sleep problems and typically developing children. Phase 2 is a randomized controlled intervention trial involving children with ASD and comorbid sleep problems, in which participants are assigned to either an aerobic exercise plus cognitive behavioral intervention group or a control group receiving cognitive behavioral strategy materials only. The intervention lasts two weeks. Outcomes related to autistic symptoms, sleep efficiency, physical activity level, attentional performance , and adaptive behaviors are assessed before and after the intervention to evaluate intervention effects.

DETAILED DESCRIPTION:
This study employs a two-phase design to investigate the effects of an acute aerobic exercise intervention combined with a parent-mediated cognitive behavioral program on sleep problems in children with Autism Spectrum Disorder (ASD). In Phase 1, cross-sectional assessments of sleep efficiency, physical fitness, and attentional performance will be conducted among children with ASD with and without sleep problems, as well as typically developing children. Phase 2 consists of a randomized intervention trial involving children with ASD and comorbid sleep problems.

During Phase 2, Eligible participants will be randomly assigned to one of two groups: (1) an acute aerobic exercise combined with cognitive behavioral intervention group, or (2) a control group receiving cognitive behavioral strategies only. The intervention period will last two weeks.

The acute aerobic exercise program will consist of moderate-to-vigorous-intensity intermittent aerobic exercise conducted twice per week, with each session lasting 30 minutes. Exercise intensity will be monitored and prescribed using standardized heart rate-based criteria to ensure participant safety and adherence to the target intensity range. Exercise sessions will be supervised by trained research staff.

The cognitive behavioral component is parent-mediated. Parents in both groups will receive structured training in cognitive behavioral strategies targeting sleep-related behaviors, including sleep routines, environmental modifications, and behavioral reinforcement techniques. Parents will be instructed to implement these strategies consistently at home on a daily basis throughout the intervention period. Adherence to the intervention will be monitored through parental reports and regular communication with the research team.

Outcome measures, including autistic symptoms, sleep efficiency, physical activity level, attentional performance and adaptive behaviors, will be assessed before and after the intervention to evaluate the effectiveness of the two intervention approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 3-11 years
2. Clinical diagnosis of Autism Spectrum Disorder and a comorbid sleep disorder
3. No diagnosis of genetic or chromosomal disorders, such as Down syndrome or Fragile X syndrome.

Exclusion Criteria:

1. Children with physical disabilities or visual or hearing impairments
2. Children who are unable to participate in vigorous physical activity due to any medical condition
3. Children with other psychiatric disorders.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency Assessed by Actigraphy | Baseline and post-intervention at Week 2
  Sleep efficiency will be calculated as the percentage of total sleep time divided by time in bed, measured using wrist-worn actigraphy.
Social Responsiveness Scale, Second Edition (SRS-2) | Baseline and post-intervention at Week 2
  Social functioning and autism-related social impairments were assessed using the Social Responsiveness Scale, Second Edition (SRS-2). The SRS-2 is a standardized, caregiver-report questionnaire designed to quantify the severity of social communication deficits and restricted and repetitive behaviors associated with autism spectrum disorder.
  The scale consists of 65 items rated on a 4-point Likert scale, with higher scores indicating greater levels of social impairment. Raw scores were converted to age- and sex-normed T-scores according to the test manual, yielding a total score and five subscale scores: Social Awareness, Social Cognition, Social Communication, Social Motivation, and Restricted Interests and Repetitive Behavior. Higher scores indicating greater severity of autism-related social impairments.
Continuous Performance Test (CPT) | Baseline and post-intervention at Week 2
  Attentional performance was assessed using the Continuous Performance Test (CPT), a computerized task designed to evaluate sustained attention and inhibitory control. During the test, children were required to respond to target stimuli and withhold responses to non-target stimuli over a continuous period of time. Key outcome measures included omission errors (failures to respond to target stimuli), commission errors (responses to non-target stimuli), reaction time, and reaction time variability, which together reflect attentional capacity, impulsivity, and response consistency.
Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) | Baseline and post-intervention at Week 2
  Adaptive functioning was assessed using the Vineland Adaptive Behavior Scales, Third Edition (Vineland-3). The Vineland-3 is a standardized caregiver-report measure designed to evaluate adaptive behaviors required for daily functioning across developmental domains.
  The assessment yields standard scores for the Adaptive Behavior Composite and domain scores for Communication, Daily Living Skills, Socialization, and Motor Skills, based on age-normed data. Higher scores indicate better adaptive functioning.
Chinese Version of the Children's Sleep Habits Questionnaire- Autism (CSHQ-Autism) | Baseline and post-intervention at Week 2
  Sleep behaviors were assessed using the Chinese version of the Children's Sleep Habits Questionnaire-Autism (CSHQ-Autism), a caregiver-reported questionnaire specifically adapted to evaluate sleep habits and sleep-related problems in children with autism spectrum disorder.
  The questionnaire consists of multiple items rated on a Likert-type scale, yielding a total sleep disturbance score and domain-specific scores reflecting common sleep difficulties, such as bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night wakings, parasomnias, sleep-disordered breathing, and daytime sleepiness. Higher scores indicate more severe sleep problems.
Repetitive Behavior Scale-Revised (RBS-R) | Baseline and post-intervention at Week 2
  Restricted and repetitive behaviors were assessed using the Repetitive Behavior Scale-Revised (RBS-R), a caregiver-reported questionnaire designed to quantify the presence and severity of repetitive and stereotyped behaviors commonly observed in individuals with autism spectrum disorder.
  The RBS-R consists of multiple items rated on a Likert-type scale, yielding a total score and subscale scores reflecting distinct domains of repetitive behavior, including Stereotyped Behavior, Self-injurious Behavior, Compulsive Behavior, Ritualistic Behavior, Sameness Behavior, and Restricted Interests. Higher scores indicate greater severity of repetitive behavior symptoms.
Chinese Version of Obstructive Sleep Apnea-18 Questionnaire (OSA-18) | Baseline and post-intervention at Week 2
  Sleep-disordered breathing-related quality of life was assessed using the Chinese version of the Obstructive Sleep Apnea-18 Questionnaire (OSA-18), a caregiver-reported instrument designed to evaluate the impact of obstructive sleep apnea symptoms on children's daily functioning and well-being.
  The questionnaire consists of 18 items rated on a Likert-type scale, yielding a total score and five domain scores: Sleep Disturbance, Physical Symptoms, Emotional Distress, Daytime Functioning, and Caregiver Concerns. Higher scores indicate greater symptom burden and poorer sleep-related quality of life.
Physical activity assessment | Baseline and post-intervention at Week 2
  Children's physical activity level was assessed using a caregiver-reported diary, which captured the frequency and duration of children's engagement in daily physical activities. This measure provided an estimate of overall physical activity participation, including total activity duration and time spent in daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- School and Graduate of Physical Therapy, Taipei, Taiwan